CLINICAL TRIAL: NCT01503996
Title: Clinical Study to Evaluate the Drinking Habits of Glaucoma Patients and Age Matched Controls
Brief Title: Drinking Habits of Glaucoma Patients and Age Matched Controls
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Dr. med., Technische Universität Dresden
Other Study IDs: Drinking/Glaucoma
Record Dates: First submitted 2011-12-01; First posted 2012-01-04 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Dehydration; Glaucoma
Keywords: dehydration; risk factor; glaucoma; Controls
MeSH Terms: conditions — Dehydration; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- glaucoma: hospitalized glaucoma patients
  Interventions: Behavioral: alter drinking habits
- controls: hospitalized patients without glaucoma
  Interventions: Behavioral: alter drinking habits

INTERVENTIONS:
Behavioral: alter drinking habits — if dehydration is apparent, more fluid intake is recommended

SUMMARY:
The purpose of this study is to examine if a chronic dehydration is a risk factor for the developement or progression of some forms of glaucoma.

DETAILED DESCRIPTION:
Glaucoma patients who are hospitalized for diurnal intraocular pressure measurements and glaucoma assessment are asked about their drinking habits. Objective evaluation of hydration status is assessed with the Body Composition Monitor (Fresenius). Retinal Vessel Analysis and Laser Doppler Flowmetry are investigated in subgroups.

The control group are also hospitalized patients who do not suffer from glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients
* controls

Exclusion Criteria:

* psychiatric disease,
* epilepsy, pregnancy,
* nutritional disorder,
* malfunction of blood clotting and wound healing,
* pacemaker,
* metallic stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients who are hospitalized for diurnal intraocular pressure measurements and glaucoma assessment.
  Controls who are hospitalizes because of an other ophthalmic disease and do not suffer from glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Dehydration | 4 years
  The composition of a patient's body, in particular a patient's water content are determined with bioimpedance spectroscopy (Body Composition Monitor, FRESENIUS)

SECONDARY OUTCOMES:
microvascular changes | 4 years
  To investigate differences in retinal vessel diameters measured with the Retinal Vessel Analyzer (RVA, IMEDOS) in glaucoma patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Pillunat, MD, Principal Investigator — University Eye Clinic Dresden
Locations (1):
- University Eye Clinic Dresden, Dresden, Germany

REFERENCES:
- [Derived] Pillunat KR, Ventzke S, Spoerl E, Furashova O, Stodtmeister R, Pillunat LE. Central retinal venous pulsation pressure in different stages of primary open-angle glaucoma. Br J Ophthalmol. 2014 Oct;98(10):1374-8. doi: 10.1136/bjophthalmol-2014-305126. Epub 2014 May 12. PMID 24820045